CLINICAL TRIAL: NCT03116503
Title: Bipolarity - Depression in Children and Adolescent Suicide Attempters: Better Diagnosis to Prevent Recurrence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 16-HPNCL-01
Record Dates: First submitted 2017-02-21; First posted 2017-04-17 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2017-04

CONDITIONS: Suicide, Attempted
Keywords: Suicide
MeSH Terms: conditions — Suicide, Attempted; Suicide

STUDY DESIGN:
Intervention Model Description: Describe the number of diagnosis of bipolar disorder and comorbid depression of suicidal behaviors in the pediatric population.
Oversight: Data Monitoring Committee: No

ARMS (1):
- bipolar disorder and comorbid depression (Experimental): number of diagnosis of bipolar disorder and comorbid depression of suicidal behaviors in the pediatric population.
  Interventions: Other: diagnosis of bipolar disorder and comorbid depression

INTERVENTIONS:
Other: diagnosis of bipolar disorder and comorbid depression — Evaluation of the number of diagnosis of bipolar disorder and comorbid depression

SUMMARY:
The purpose of the study is to describe the number of diagnosis of bipolar depression and comorbid suicidal behavior according to the diagnostic criteria of the DSM-5.

DETAILED DESCRIPTION:
This study is a prospective, routine care, covering pediatric population suicidal (who attempted suicide) and suicide (with suicidal ideas with planning) hospitalized in the pediatric hospital in Nice- Lenval Hospital.

The main objective of the study is to describe the number of diagnosis of bipolar depression and comorbid suicidal behavior according to the diagnostic criteria of the DSM-5.

The secondary objectives are: 1) comparison of the suicide attempt rate of recurrence at 6 months and 12 months among subjects with a diagnosis of mood disorder (depression or bipolar) and subjects with a diagnosis mood disorder; 2) the identification of specific suicidal recurrence risk factors in the diagnosis of mood disorder; 3) comparing the diagnostic evaluation field (ICD-10 criteria) vs standardized assessment (DSM-5 criteria).

For this the investigator propose an observational cohort study, single center, on a trailing 12 months after inclusion.

The topics are selected and included consecutively over a period of 12 months. The inclusion criteria are: 1) children - teenagers age: 6-18 years inclusive; 2) hospitalization for suicide attempt or suicidal ideation with planning in the Pediatric Hospital of Nice Lenval Hospital; 3) French patients; 4) speaking parents 5) affiliation to the social security system.

The criterion for inclusion is not the refusal or failure to realize the Kiddie - SADS with the subject and / or his parents.

The number of subjects to be included is estimated at 100. At baseline: standardized assessment of comorbid psychiatric diagnosis according to DSM-5 Mood disorders according to DSM-IV R criteria for other diagnoses. The investigatorwill use the KIDDIE-SADS, semi-structured interview for diagnostic purposes adapted to the DSM for that assessment.

The patients were distributed into two groups: mood disorder group - group without mood disorder.

In parallel, the field team evaluates blind psychiatric diagnosis according to ICD-10 criteria.

The population included subjects is described: clinicaly - demographic - overall operation - individual and family psychiatric history.

The topics included are reassessed at 6 months and 12 months. At 6 months: occurrence of an attempted suicide or recurrence of suicidal thoughts with planning - overall operation - clinical condition. At 12 months: re standardized diagnostic evaluation with KIDDIE-SADS and re identical clinical evaluation at 6 months.

The recidivism risk factors and recidivism rates are evaluated in both groups. The primary endpoint of the study is the attempt recurrence rate of suicide.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized at Fondation Lenval/ pediatric hospital of Nice-CHU Lenval for suicide attempt and / or suicidal ideas with planning
* French-speaking patient
* Francophone parents
* Affiliation to asocial security system

Exclusion Criteria:

* Refusal or impossibility of carrying out the KIDDIE-SADS questionnaire

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
diagnosis of bipolar disorder and comorbid depression | At baseline during inclusion visit
  Describe the number of diagnosis of bipolar disorder and comorbid depression of suicidal behaviors in the pediatric population.

SECONDARY OUTCOMES:
recurrence rates | comparison between 6 month and 12 month
  compare the recurrence rates at 6 and 12 months between bipolar and depressed patients and patients not diagnosed with a mood disorder
risk factors for suicidal recidivism | At baseline during inclusion visit
  To compare the risk factors for suicidal recidivism between bipolar and depressed patients
comorbid diagnoses | At baseline during inclusion visit
  Compare the comorbid diagnoses obtained by the standardized assessment (Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) for mood disorders and DSM-IVR for other diagnoses) vs. field assessment (CIM-10) (Classification internationale des maladies-10)

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie DUGAND, MD, Principal Investigator — Fondation Lenval
Locations (1):
- Fondation Lenval, Hôpitaux pédiatriques de Nice CHU Lenval, Nice, France

IPD SHARING:
Plan to Share IPD: No